CLINICAL TRIAL: NCT07216976
Title: Adaptive DBS Algorithm for Personalized Therapy in Parkinson's Disease (ADAPT-PD) China Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT 24043
Record Dates: First submitted 2025-10-09; First posted 2025-10-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single-arm who received aDBS "Best" Mode (Dual or Single Threshold ) (Experimental)
  Interventions: Device: Percept™ PC with Adaptive DBS (aDBS™)

INTERVENTIONS:
Device: Percept™ PC with Adaptive DBS (aDBS™) — Subjects for whom meet the LFP screening criteria and can be acceptably configured on the "Best" aDBS mode (Dual or Single Threshold) will receive "Best" Mode aDBS treatment and enter the aDBS Evaluation Phase.
  Other Names: aDBS

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the Medtronic Percept PC with Adaptive DBS therapy (aDBS) for Parkinson's Disease in China.

The main question it aims to answer is: To demonstrate at least 50% of subjects meet a success criterion relative to stable cDBS.

DETAILED DESCRIPTION:
The ADAPT-PD China Study will utilize both Dual and Single Threshold aDBS modes (algorithms). Prospective, multicenter, open label comparison (with single-blind aDBS mode from aDBS randomization to evaluation phase), single arm clinical trial designed to evaluate the effectiveness of the Medtronic Percept PC INS with aDBS for Parkinson's Disease in China.

The study is expected to be conducted at approximately 5 centers located in China.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet all general inclusion/exclusion criteria (as assessed at the Enrollment Visit)
2. Subjects must meet the LFP screening inclusion criterion (as assessed at the LFP Screening Visit)

General (Assessed at Enrollment Visit):

1. Subject has idiopathic Parkinson's disease
2. Subject is implanted (>3 months prior to enrollment for new INS implants or >1 month from INS replacement) with Percept PC (Model B35200) and Medtronic DBS leads (Model 3387, 3389, B33005 or B33015) and extensions (Model 37086 or B34000) bilaterally in the same target (physician confirmed), STN or GPi
3. In the opinion of the investigator, the subject responds to DBS Therapy.
4. Based on the opinion of the investigator, the subject's cDBS parameters and PD medications are stable (no changes within the last 4 weeks) and expected to remain stable from enrollment through the end of the aDBS Evaluation Phase
5. Subject is configured to monopolar or dual monopolar stimulation using contacts 1 and/or 2 (9 and/or 10) on at least one side
6. Subject is willing and able to attend all study-required visits and complete the study procedures (e.g. 1-month recall questionnaires, MDS-UPDRS III, Off stim/Off med visit)
7. Subject (or legally authorized representative) has the ability to understand and provide written informed consent for participation in the study prior to the study-related procedures being conducted
8. Subject is a male or non-pregnant female. If female of child-bearing potential, and if sexually active, must be using, or agree to use, a medically-acceptable method of birth control as confirmed by the investigator

LFP Screening Inclusion Criteria (Conducted during LFP Screening Visit):

1. Subject has Alpha - Beta band (8-30 Hz) amplitude ≥ 1.2 μVp detected on either left and/or right DBS leads on sensing channels 0-2, 0-3, 1-3, 8-10, 8-11, or 9-11.

Exclusion Criteria:

General (Assessed at the Enrollment Visit):

1. Subject and/or caregiver is unable to utilize the patient programmer
2. Subject has more than one lead in each hemisphere of the brain
3. Subject has cortical leads or additional unapproved hardware implanted in the brain
4. Subject has more than one INS
5. At enrollment, the subject's INS has a predicted battery life of <1 year
6. Subject has Beck Depression Inventory II (BDI-II)>25
7. Subject requires diathermy, transcranial magnetic stimulation (TMS), or electroconvulsive therapy (ECT)
8. Subject has a metallic implant in the head, (e.g., aneurysm clip, cochlear implant)
9. Subject has, or plans to obtain, an implanted electrical stimulation medical device anywhere in the body (e.g., cardiac pacemaker, defibrillator, spinal cord stimulator)
10. Subject has, or plans to obtain, an implanted medication pump for the treatment of Parkinson's disease (e.g., DUOPATM infusion pump) and/or portable infusion pump
11. Based on the opinion of the investigator, the subject has an abnormal neurological examination that would preclude them from study participation
12. Subject is breast feeding
13. Subject is under the age of 18 years
14. Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound the results of this study as determined by the Medtronic study team
15. Subjects with signal artifact on all 6 aDBS sense pathways (3 each on both DBS leads) which preclude the clinician from setting thresholds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
"On" time without troublesome dyskinesia (i.e. Good "On" Time) | From the cDBS baseline to aDBS evaulation phase at about 1 month
  Proportion of aDBS subjects meet a success criterion relative to stable cDBS.The success criterion: no worse than 2 hours/day less of "On" time without troublesome dyskinesia (i.e. Good "On" Time) during aDBS compared to cDBS.

OTHER OUTCOMES:
Assess the Adverse Event among the Participants | From enrollment to the end of treatment at around 12 months to 17.5 months
  To characterize:
  * Stimulation-related adverse events (AEs)
  * Adverse events including serious adverse events (SAEs) and device deficiencies

CONTACTS AND LOCATIONS:
Overall Officials: Alex Xie, Clinical Research&Medical Science Director, Study Director — Medtronic (Shanghai) Management Co. Ltd.
Locations (5):
- China (5):
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Hospital, Guangzhou, Guangdong
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
Due to the personal data protection, the IPD for each site will only be used for this study purpose and will only be opened for site investigators. Also, the informed consent doesn't include sharing IPD with other researchers.